CLINICAL TRIAL: NCT01026363
Title: hCAP18 Levels and Vitamin D Deficiency in Chronic Kidney Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Kidney Foundation, United States (Other)
Responsible Party: Principal Investigator, Ishir Bhan, MD, MPH, Assistant in Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-P-001050/1; 1K23DK081677 (NIH)
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Kidney Disease; Vitamin D Deficiency
Keywords: Vitamin D; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Vitamin D Deficiency | interventions — Ergocalciferols; Vitamin D; Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ergocalciferol (Experimental): Ergocalciferol intervention arm
  Interventions: Drug: Ergocalciferol
- calcitriol (Experimental): calcitriol intervention arm
  Interventions: Drug: Calcitriol

INTERVENTIONS:
Drug: Ergocalciferol — Ergocalciferol 50,000 IU capsule, one dose every other day x 5 doses
  Other Names: Vitamin D
  Arms: ergocalciferol
Drug: Calcitriol — 0.25 mcg tablet once daily for 14 days
  Other Names: vitamin d
  Arms: calcitriol

SUMMARY:
The human immune system produces a protein called hCAP18 (also known as LL-37 or cathelicidin). This protein is believed to help the body to fight infections. Studies suggest that vitamin D may important in the production of hCAP18. This study is designed to test the ability of two different forms of vitamin D to affect levels of hCAP18. Vitamin D and hCAP18 levels will be measured during an initial visit. Individuals who are vitamin D deficient will be randomly assigned to receive one of two forms of vitamin D for two weeks. After this, follow-up levels will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Chronic Kidney Disease stage 3-4 (estimated glomerular filtration rate 15-60 ml/min)

Exclusion Criteria:

* 6 month history of hypercalcemia, hyperphosphatemia, or nephrolithiasis
* use of active vitamin D analog within 30 days
* functioning renal transplant
* Symptoms of active infection
* Granulomatous disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
hCAP18 levels | 2 weeks

SECONDARY OUTCOMES:
1,25-dihydroxyvitamin D | 2 weeks
25-hydroxyvitamin D | 2 weeks
calcium | 2 weeks
phosphorus | 2 weeks
Parathyroid hormone | 2 weeks
T-cell subsets | 2 weeks
  Measures of different types of T-cells

CONTACTS AND LOCATIONS:
Overall Officials: Ishir Bhan, MD MPH, Principal Investigator — Massachusetts General Hospital, Massachusetts Institute of Technology
Locations (1):
- Massachusetts Institute of Technology, Cambridge, Massachusetts, United States

REFERENCES:
- [Background] Gombart AF, Bhan I, Borregaard N, Tamez H, Camargo CA Jr, Koeffler HP, Thadhani R. Low plasma level of cathelicidin antimicrobial peptide (hCAP18) predicts increased infectious disease mortality in patients undergoing hemodialysis. Clin Infect Dis. 2009 Feb 15;48(4):418-24. doi: 10.1086/596314. PMID 19133797